CLINICAL TRIAL: NCT05892120
Title: The Effectiveness of a Smartphone App on Medication Adherence and Psychotic Symptoms and Cognitive Functions in Patients With Schizophrenia
Brief Title: A Smartphone App on Medication Adherence
Acronym: App
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMURCT20200096
Record Dates: First submitted 2023-05-16; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Medication Adherence
Keywords: schizophrenia; medication adherence; smartphone app; psychiatric symptoms
MeSH Terms: conditions — Medication Adherence; Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: The control group only received usual care, the PANSS and MMSE were used to assess psychiatric symptoms and cognitive functions before (week 0) and after 8 weeks.
- experimental group: The experimental group use the MedAdhere app for eight weeks, the PANSS and MMSE were used to assess psychiatric symptoms and cognitive functions before (week 0) and after (week 8) intervention.
  Interventions: Behavioral: the MedAdhere app

INTERVENTIONS:
Behavioral: the MedAdhere app — The experimental group downloaded and used the MedAdhere app on their personal smartphones during this 8-week study
  Groups: experimental group

SUMMARY:
This is an experimental study which aims to explore the effectiveness of a smartphone app for medication adherence (MedAdhere app) among schizophrenic patients for eight weeks.

DETAILED DESCRIPTION:
Schizophrenia is a mental disorder that causes severe functional disabilities and imposes a heavy economic burden. Poor medication adherence is one of the major causes of relapse of psychiatric symptoms in schizophrenic patients. This is an experimental study which aims to explore the effectiveness of a smartphone app for medication adherence (MedAdhere app) among schizophrenic patients for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia
* aged 20 to 65 years
* able to read traditional Chinese
* owning a smartphone
* currently admitted at a psychiatric day-care center

Exclusion Criteria:

* Intellectually disabled or severe cognitive function impairment (Dementia)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Schizophrenia is a brain disorder that is possibly related to the reduction of neural connections in the prefrontal cortex or imbalances in dopaminergic neurons in brain. It can be induced by genetic, social, physiological, psychological, and other factors, resulting in cognitive, emotional, behavioural, and perception dysfunction.
  At present, new generations of anti-psychotic drugs have become available, allow patients to stabilise their condition with less side effect by receiving regular drug treatment. However, medication non-adherence can cause disorder progression, compromise the patient's quality of life, and increase medical expenses
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-07-25 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
psychiatric symptoms | Change from Baseline psychiatric symptoms at 8 weeks
  The positive and negative syndrome scale was used to measure participants' psychiatric symptoms.
  Of the 30 items on the scale, seven are positive symptoms, seven are negative symptoms, and 16 are general psychopathology symptoms. Symptom severity for each item is rated according to the anchoring points in the 7-point scale (1 = absent; 7 = extreme) that best describe the symptom (Kay et al., 1987). The PANSS score is the sum of ratings across items, ranging from 7 to 49 for the Positive, Negative Scales, and 16 to 112 and 16 to 112 for the General Psychopathology Scale.
cognitive functions | Change from Baseline cognitive functions at 8 weeks
  The Mini-Mental State Examination was used to measure participants' cognitive functions.
  The MMSE consists of 15 questions for assessing the following seven cognitive domains: orientation in time and place, memory registration and recall, attention and calculation, and language. The total MMSE score ranged from 0 to 30, and higher scores indicate better cognitive functions.
Medication adherence rate | Change from Baseline Medication adherence' rate at 8 weeks
  Utilizing cloud-based platforms to compute the medication adherence rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen HH, Hsu HT, Lin PC, Chen CY, Hsieh HF, Ko CH. Efficacy of a Smartphone App in Enhancing Medication Adherence and Accuracy in Individuals With Schizophrenia During the COVID-19 Pandemic: Randomized Controlled Trial. JMIR Ment Health. 2023 Dec 14;10:e50806. doi: 10.2196/50806. PMID 38096017